CLINICAL TRIAL: NCT00066417
Title: Pilot Study Of T-Cell-Depleted Peripheral Blood Stem Cell Transplantation From Partially Matched Related Donors For Patients With High-Risk Leukemia
Brief Title: Peripheral Stem Cell Transplant in Treating Patients With High-Risk Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was withdrawn for drug availability issues.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000315900; NHLBI-03-H-0209; NCT00062725 (obsolete NCT alias)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2006-11

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Myelodysplastic/Myeloproliferative Diseases
Keywords: essential thrombocythemia; polycythemia vera; blastic phase chronic myelogenous leukemia; secondary myelodysplastic syndromes; previously treated myelodysplastic syndromes; adult acute myeloid leukemia in remission; childhood acute myeloid leukemia in remission; de novo myelodysplastic syndromes; secondary acute myeloid leukemia; accelerated phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent adult acute myeloid leukemia; relapsing chronic myelogenous leukemia; recurrent childhood acute myeloid leukemia; chronic idiopathic myelofibrosis; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Myelodysplastic-Myeloproliferative Diseases; Thrombocythemia, Essential; Polycythemia Vera; Blast Crisis; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Acute; Primary Myelofibrosis; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Congenital Abnormalities | interventions — Cyclophosphamide; Cyclosporine; fludarabine phosphate; Methylprednisolone; Thiotepa; Biological Therapy; Bone Marrow Transplantation; Drug Therapy; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: methylprednisolone
Drug: therapeutic allogeneic lymphocytes
Drug: thiotepa
Procedure: allogeneic bone marrow transplantation
Procedure: biological therapy
Procedure: bone marrow ablation with stem cell support
Procedure: bone marrow transplantation
Procedure: chemotherapy
Procedure: leukocyte therapy
Procedure: non-specific immune-modulator therapy
Procedure: peripheral blood lymphocyte therapy
Procedure: peripheral blood stem cell transplantation
Procedure: radiation therapy

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor peripheral stem cell transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the stem cells from a related donor, that do not exactly match the patient's blood, are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

PURPOSE: This phase II trial is studying how well peripheral stem cell transplant works in treating patients with high-risk leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of a preparative regimen comprising total body irradiation, cyclophosphamide, thiotepa, and fludarabine, but without anti-thymocyte globulin, in patients with high-risk leukemia treated with peripheral blood stem cell transplantation from partially matched related donors.
* Determine the incidence of graft failure, acute graft-versus-host disease (GVHD), and treatment-related mortality in patients treated with this regimen.
* Determine rates of chronic GVHD and relapse in patients treated with this regimen.
* Determine disease-free and overall survival in patients treated with this regimen.

OUTLINE: This is a pilot study.

Patients receive a preparative regimen comprising total lymphoid irradiation once daily on days -13 to -11; cyclophosphamide IV over 1 hour on days -8 and -7; thiotepa IV over 4 hours every 12 hours on day -6; fludarabine IV over 30 minutes on days -5 to -1; and total body irradiation once on day -1. Patients also receive cyclosporine IV over 12 hours on days -8 to -1 and methylprednisolone IV twice daily on days -3 and -2. Patients receive CD34-enriched T-cell-depleted allogeneic stem cell infusion on day 0.

Patients with disease progression or uncontrolled infection but without grade II or greater graft-versus-host disease may receive up to 3 donor lymphocyte infusions at least 4 weeks apart until disease regression.

Patients are followed at least weekly until day 100 and then at 6, 12, 18, 24, 36, and 48 months.

PROJECTED ACCRUAL: A total of 20-51 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * High-risk myelodysplastic syndromes (MDS), meeting 1 of the following criteria:

    * Transformation to acute leukemia defined by at least 15% blasts
    * Secondary to prior treatment with chemotherapy and/or radiotherapy
    * Presence of complex cytogenetics (at least 3 karyotypic abnormalities)
    * Monosomy or deletion of chromosome 7
  * Acute myeloid leukemia (AML), meeting 1 of the following criteria :

    * High-risk AML in first remission and meeting 1 of the following criteria:

      * At least 3 karyotypic abnormalities
      * Monosomy or deletion of chromosome 5 or 7 = 11q23 chromosomal abnormality
      * Prior diagnosis of MDS
      * Received prior radiotherapy or chemotherapy
    * In second or subsequent remission
    * Primary induction failure or partial remission
    * Untested or sensitive relapse
  * Chronic myelogenous leukemia, meeting 1 of the following criteria:

    * Blast crisis
    * Accelerated phase disease that has failed prior treatment with imatinib mesylate, defined as a failure to achieve hematologic response after 3 months of standard dose (600 mg/day) therapy or disease progression on therapy
  * Myeloproliferative disease

    * The following diagnoses are eligible:

      * Agnogenic myeloid metaplasia
      * Essential thrombocythemia
      * Polycythemia vera
    * Must have evidence of transformation to acute leukemia
  * Acute lymphocytic leukemia (ALL), meeting 1 of the following criteria:

    * High-risk ALL in first remission defined by 1 of the following:

      * t(9;22) or 11q23 chromosomal abnormality
      * Complete response at least 4 weeks after induction therapy OR requiring at least 2 induction regimens
    * Second or subsequent remission
* No relapsed leukemia refractory to appropriate salvage therapy
* Availability of an HLA-mismatched family donor

  * Donor age 75 or under
* No better donor alternative (i.e., HLA-matched related or unrelated stem cell donor) is available

PATIENT CHARACTERISTICS:

Age

* 10 to 50

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin no greater than 4 mg/dL
* Transaminases no greater than 3 times upper limit of normal

Renal

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* LVEF at least 40%

Pulmonary

* DLCO at least 65% of predicted

Other

* Not pregnant
* Negative pregnancy test
* HIV negative
* No other prior malignancy except basal cell or squamous cell skin cancer or a remote history of cancer now considered cured
* No major organ dysfunction that would preclude transplantation
* No major anticipated illness or organ failure that would preclude transplantation
* No severe psychiatric illness or mental deficiency that would preclude giving informed consent or complying with study
* No uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Estimated)
Dates: Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Incidence of graft failure 100 days post-transplant
Incidence of acute and chronic graft-vs-host disease100 days post-transplant
Transplant-related mortality 100 days post-transplant
Disease-free survival 100 days post-transplant
Overall survival 100 days post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Bipin N. Savani, MD, Study Chair — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- NIH - Warren Grant Magnuson Clinical Center, Bethesda, Maryland, United States